CLINICAL TRIAL: NCT01066260
Title: Efficacy of a Probiotic Formulation on Energy Balance in Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-24 MET
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Probiotics; Energy balance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental)
  Interventions: Dietary Supplement: Probiotic formulation
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic formulation — Twice a day for 24 days
  Arms: Probiotic
Other: Placebo — Twice a day for 24 days
  Arms: Placebo

SUMMARY:
Probiotic administration is associated with health benefits on gut barrier integrity and immunological functions of the gastrointestinal tract. Recently, probiotic consumption was proposed to reduce fat mass and body weight in rodents (Lee HY. et al. 2006; Hamad EM. et al. 2009). Changes in energy metabolism might be involved in the effects of probiotics on weight control.

The objective of this study was to assess the efficacy of the consumption of a probiotic formulation on energy balance in overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Masss Index (BMI) 25 - 30 kg/m2
* Healthy (determined by medical questionnaire)
* Able to commit to the duration of the study
* Providing consent for participation

Exclusion Criteria:

* History of cardiovascular disease (CVD), diabetes, cancer, renal, thyroid or hepatic disease
* History of gastrointestinal surgery
* History of sleep disorders
* Recent bacterial infection (< 2 weeks)
* Weight loss > 5 kg in the last 3 months
* Under antibiotics or treatments (medical or nutritional program) affecting body weight, appetite, energy expenditure lipid-lowering, hypertension or inflammation or glucose control for the last 3 months or taking hormone replacement therapy
* Excessive consumption of products enriched in probiotics (> 4 servings per week) within the last 4 weeks before the start of the study
* History of drug or alcohol abuse (> 2 drinks daily)
* Regular smokers (more than 5 cigarettes a day)
* Not eating breakfast regularly or eating breakfast before 6h00.
* Not willing to eat any of the foods to be served in the study for any reason
* Physical activity level > 150 min of moderate or intense exercise per week
* Concurrent or recent intervention study (within 60 days)

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Energy intake | Lunch

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD, Principal Investigator — Société des Produits Nestlé (SPN)
Locations (1):
- Nestlé Research Center, Lausanne, Canton of Vaud, Switzerland